CLINICAL TRIAL: NCT01077349
Title: Early Continuous High Volume Veno-venous Hemofiltration vs. Standard Care for Post-cardiac Surgery Shock Requiring High Doses Catecholamines. The HEROICS Study: HEmofiltration to Rescue Severe shOck followIng Cardiac Surgery
Brief Title: High Volume Veno-venous Hemofiltration Versus Standard Care for Post-cardiac Surgery Shock
Acronym: HEROICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071223
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2012-10

CONDITIONS: Shock
Keywords: Cardiac surgery; Shock; Continuous Veno-Venous Haemofiltration; Continuous Renal Replacement Therapy; Renal Insufficiency; Acute
MeSH Terms: conditions — Shock; Renal Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high volume hemofiltration (Experimental)
  Interventions: Procedure: high volume hemofiltration
- standard care (Active Comparator)
  Interventions: Procedure: standard care

INTERVENTIONS:
Procedure: high volume hemofiltration — (80 ml/kg/h or a maximum of 8L/h) for 48 hours following heart surgery. Hemofiltration will be stopped after 48h if diuresis >1500 ml without diuretics and if IV infusion of catecholamines is less than 0.1 microg/kg/min of epinephrine, 0.2 microg/kg/min of norepinephrine or the sum of epinephrine + nor epinephrine/2 is less than 0.1 microg/kg/min. In other cases, hemodiafiltration (CVVHDF) will be initiated until the above objectives are reached, with equal flow rate of dialysate and reinfusion fluid, the sum of which being <35 ml/kg/h (or a maximum of 3500 ml/h).
  Arms: high volume hemofiltration
Procedure: standard care — extra-renal replacement therapy (CVVHDF mode, total effluent <35 ml/kg/h or a maximum of 3500 ml/h) will be initiated only if the following criteria are met:
  * Serum creatinine > 350 micromol/L or increase x3.0 from pre-operative value OR
  * Diuresis < 0.3 ml/kg/h for 24 hours despite adequate fluid resuscitation OR
  * Or serum urea > 36 mmol/l OR
  * Or life threatening hyperkalemia
  Arms: standard care

SUMMARY:
This study seeks to determine if early continuous High Volume Veno-venous Hemofiltration (HVHF) reduces 30-day all cause mortality in post-cardiac surgery patients developing shock requiring high doses catecholamines.

DETAILED DESCRIPTION:
Study Title - Early continuous high volume veno-venous hemofiltration vs. standard care for post-cardiac surgery shock requiring high dose catecholamines. An open label randomized multicenter controlled trial. The HEROICS Study: HEmofiltration to Rescue severe shOck followIng Cardiac Surgery.

Clinical Phase - III Study Rationale - Systemic inflammatory response syndrome associated with cardiac surgery under cardiopulmonary bypass (CPB) shares many pathophysiologic features of septic shock and post-resuscitation syndrome. Since high volume hemofiltration has been shown to markedly improve hemodynamic profile and survival in these situations, there is a strong rationale for testing, with an adequately powered randomized controlled trial, this purification technique in patients developing post-cardiac surgery shock requiring high doses catecholamine.

Trial Design -

The proposed study will compare high volume hemofiltration (80 ml/kg/h or a maximum of 8L/h) for 48 hours following heart surgery to standard treatment, where extra-renal replacement therapy (CVVHDF mode, total effluent <35 ml/kg/h) will be initiated only if the following criteria are met:

* Serum creatinine > 350 micromol/L or increase x3.0 from pre-operative value OR
* Diuresis < 0.3 ml/kg/h for 24 hours despite adequate fluid resuscitation OR
* Or serum urea > 36 mmol/l OR
* Or life threatening hyperkalemia. In the experimental arm, hemofiltration will be stopped after 48h if diuresis >1500 ml without diuretics and if IV infusion of catecholamines is less than 0.1 microg/kg/min of epinephrine, 0.2 microg/kg/min of norepinephrine or the sum of epinephrine + norepinephrine/2 is less than 0.1 microg/kg/min. In other cases, hemodiafiltration (CVVHDF) will be initiated until the above objectives are reached, with equal flow rate of dialysate and reinfusion fluid, the sum of which being 35 ml/kg/h (or a maximum of 3500 ml/h).

Subject Participation - 90 days

Rationale for Number of Subjects - The study will follow a sequential analytical plan with stopping rules based on the triangular test. The expected mortality of the control group is expected to be 25% and the expected absolute mortality reduction with the experimental treatment of 12%. For 80% power and a 5% α-risk, the study characteristics, calculated with the triangular test, are as follows: a maximum of 540 subjects to be included and a 90% probability of stopping the study before 330 subjects have been included. With an inclusion rate of 120-150 patients per year, the maximum duration of the study is 2 years and 3 months and the probability of stopping the study before 18 months is 90%.

Approximate duration of Study - 27 months

Study Objective(s) Primary - The primary study outcome is death from all causes at 30 days after randomisation.

Secondary

1. Mortality 60 and 90 days following study enrollment
2. ICU and Hospital mortality
3. Mortality adjusted on the type of surgery and patient severity at randomization
4. Duration of catecholamine infusion and number of catecholamine-free days at 30 days following study enrollment
5. Duration of renal replacement therapy and number of renal replacement therapy -free days at 30 days following study enrollment
6. Recovery of renal failure and dialysis independent survival
7. Duration of mechanical ventilation and number of mechanical ventilation -free days at 30 days following study enrollment
8. SOFA score on days 1, 2 ,3 ,4 ,7 ,15 , and 30 following study enrollment
9. Reduction in markers of overt coagulation and inflammation at days 2, 4 and 7 following study enrollment
10. ICU and Hospital length of stay
11. Mortality analysis according to subgroups of patients (type of surgery, severity at randomization, renal function at randomization)

Approximate Number of Subjects - 330

Approximate Number of Study Centres - 8 centres distributed in France will participate in the study.

Treatment Administration - Each participant will be randomised to receive high volume hemofiltration (CVVH, 80 ml/kg/h or a maximum of 8L/h) for 48 hours following heart surgery or standard treatment, where extra-renal replacement therapy (CVVHDF mode, total effluent <35 ml/kg/h) will be initiated only if criteria for renal failure are met.

Safety Evaluation - Safety for individual patients will be assessed on an ongoing basis by physical examination, including vital signs, outputs from dialysis machine records, laboratory assessments, and monitoring of adverse events. Overall study safety will be ensured by an Independent Data Safety Monitoring Committee, independent from all Trial investigators, which will perform ongoing review of predefined safety parameters and study conduct.

Efficacy Evaluation - Overall survival at 30 days post randomisation

Statistical Analysis - The first analysis is scheduled after the inclusion of 60 subjects. Thereafter, stopping rules are scheduled to be sequentially applied, based on the triangular test. This will allow us to stop the trial as soon as there are sufficient evidence that one of the 2 treatment strategies are more dangerous or that there was no longer a chance of demonstrating the postulated treatment difference of 12%, while controlling the risks of type I and II errors. Sequential analyses will be conducted every 20 patients. The baseline and outcome variables will be compared using Students t test, Chi squared and the Mann-Whitney U test as appropriate. Kaplan-Meier survival curves for the 30 days following randomization will be compared with a log-rank test., with survival being calculated from the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac surgery with cardiopulmonary bypass
2. Patient still on high doses catecholamines 3 to 24 hours following cardiac-surgical ICU admission. High doses catecholamines is defined by IV infusion of :

   1. Epinephrine >0.2 microg/kg/min or
   2. Norepinephrine >0.4 microg/kg/min or
   3. Epinephrine + (Norepinephrine /2) >0.2 microg/kg/min
   4. Cardiac assistance using ECMO/ECLS technique are considered equivalent to high doses catecholamines.
3. Informed consent has been obtained from next of kin or when consent cannot be obtained, the intervention is randomized, and written informed consent obtained from the patient as soon as he regains consciousness. This practice is consistent with the French law for clinical research.

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. Chronic hemodialysis prior to heart surgery
4. Body weight >120 kg
5. Moribund state, defined as SAPS 2 score> 90
6. Severe underlying disease with survival expectancy of less than 8 days
7. Decision to withhold or withdraw active therapeutics
8. PrismaFlex machine unavailable in the unit
9. Intravascular access with dialysis catheter impossible -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Death from all causes at 30 days after randomisation | 30 days

SECONDARY OUTCOMES:
Mortality 60 days following study enrollment | 60 days
ICU mortality | 90 days
Mortality adjusted on the type of surgery and patient severity at randomization | 90 days
Mortality 90 days following study enrollment | 90 days
Hospital mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Alain Combes, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Result] Combes A, Brechot N, Amour J, Cozic N, Lebreton G, Guidon C, Zogheib E, Thiranos JC, Rigal JC, Bastien O, Benhaoua H, Abry B, Ouattara A, Trouillet JL, Mallet A, Chastre J, Leprince P, Luyt CE. Early High-Volume Hemofiltration versus Standard Care for Post-Cardiac Surgery Shock. The HEROICS Study. Am J Respir Crit Care Med. 2015 Nov 15;192(10):1179-90. doi: 10.1164/rccm.201503-0516OC. PMID 26167637
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787